CLINICAL TRIAL: NCT02590952
Title: An Open-label, Multi-Centered, Dose Escalation Phase Ib Study (Expansion Stage) of Epitinib (HMPL-813) in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of Epitinib(HMPL-813) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-813-00CH1
Record Dates: First submitted 2013-10-14; First posted 2015-10-29 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2019-02

CONDITIONS: Solid Tumor
Keywords: safety, PK

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epitinib (Experimental): Epitinib is a capsule in the form of 5mg,20 mg, and 40 mg. Route: oral (daily)
  Interventions: Drug: Epitinib

INTERVENTIONS:
Drug: Epitinib — The starting daily dose is 20 mg. Dose escalation will follow daily dose of 40 mg,80 mg, 120 mg, 160 mg, 200 mg, and 250 mg. A 3+3 design applies to this study. Patients will continue taking Epitinib until they experience intolerable adverse events or their diseases are confirmed to be progressed.
  Other Names: HMPL-813

SUMMARY:
Epitinib (HMPL-813) is a selective EGFR tyrosine kinase inhibitor. Epitinib has demonstrated strong inhibitory effects on multiple tumors with overexpressed EGFR or sensitive EGFR mutations in pre-clinical setting. This first-in-human study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity(DLT), safety and tolerability, pharmacokinetics (PK), and preliminary anti-tumor activity of Epitinib.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology confirmed solid tumors
* Failed to standard treatment or no standard treatments for uncontrolled, recurrent and/or metastatic advance tumor (whatever previous surgery conditions)
* Age 18-70
* ECOG 0-2, and no worse within 7days
* Life expected > 12 weeks
* written informed consent form voluntarily
* For dose expansion cohort, subjects must be eligible for the following inclusion criteria:
* EGFR sensitizing mutation in exon 19 deletion or exon 21(L858R).
* Histologically or cytologically confirmed advanced NSCLC with brain metastasis. No prior brain radiotherapy or brain metastasis progressed after brain radiotherapy delivered assessed by RECIST 1.1.
* No prior EGFR-TKI treatment. Or subjects who treated with EGFR-TKI developed brain lesions during EGFR-TKI therapy or the existing brain lesions progressed but with stable extra-cranial lesions.
* Treatment failure of prior systemic chemotherapy for locally advanced or metastasized NSCLC or intolerance to chemotherapy. Or subjects with disease relapse after treated with adjuvant or neo-adjuvant chemotherapy.
* With at least one measurable disease ( RECIST 1.1).

Exclusion Criteria:

* Lab testing within 2 weeks before enrolled, AND ANC<1.5×10 9/L, platelet<75×10 9/L, or Hb<9g/dL,
* Serum Total Bilirubins > ULN, ALT/AST≥ULN without liver metastasis, or ALT/AST≥2.5ULN with liver metastasis
* Serum creatinine >1.5ULN or creatinine clearance <40ml/min
* Diastolic systolic pressure≥140mmHg or systolic diastolic pressure≥90mmHg whatever anti-hypertension drug used,
* Serum potassium <4.0mmol/L(whenever potassium implemented), serum calcium(ionic or albumin-type calcium) or serum magnesium outside normal ranges(whenever implemented)
* Within previous 4 weeks treated by systemic anti-tumor therapy, or radiotherapy, immune therapy, biological or hormonal therapy, and clinical trials.
* Unrecovered from any previous therapy related toxicity to CTCAE 0 or 1or unrecovered from any previous surgery
* Known dysphagia or drug malabsorption
* Active infections such as acute pneumonia, hepatitis B immune-active periodphase
* ocular surface diseases or dry eye syndrome
* skin disease with obvious symptoms and signs
* significant cardiovascular disease, including II-IV atrioventricular block, and acute myocardial infarction within 6 months, significant angina or Coronary artery bypass graft within 6 months
* Female patients who are pregnant or feeding, or childbearing potential patient with pregnant testing positive
* Any abnormal of clinical and laboratory so that patients unsuitable to attend the trial sine in the opinion of the investigator
* Patients unable to comply with the protocol since significant psychological or psychogenic abnormal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
incidence of all types/grades of adverse events | from first patient in till 30 days after the last patient last visit. It is estimated that last patient last visit happens in Oct 2016.
  for each patient, adverse events are collected from the date of consent until 30 days after trial discontinuation

SECONDARY OUTCOMES:
Objective Response Rate | An average of one year
Area under the plasma concentration versus time curve (AUC) | At single-dose stage (day 1-day 7): predose, 0.5,1, 2, 3, 4, 5, 6, 8,12,24, 36, 48, 72, 144 hours post-dose.
  Based on single-dose PK result, multi-dose stage subjects take epitinib either once a day or twice a day. For twice a day epitinib uptake, on day 1/14/28, PK samples are collected predose, 1, 4, 8, 12 hours post-dose in the morning and 4 hours post-dose in the evening. On day 2/3/7, PK samples are collected predose, 4, 12 hours post-dose in the morning and 4 hours post-dose in the evening. On day 15/29/56, PK samples are collected predose in the morning.
  For once a day epitinib uptake, on day 1/14/28 PK samples are collected predose, 0.5, 1, 2, 4, 6, 8, 12 hours post-dose. On day 7, PK samples are collected predose and 4 hours post-dose. On day 2/15/29/56, PK samples are collected predose in the morning.
Peak Plasma Concentration (Cmax) | At single-dose stage (day 1-day 7): predose, 0.5,1, 2, 3, 4, 5, 6, 8,12,24, 36, 48, 72, 144 hours post-dose.
  Based on single-dose PK result, multi-dose stage subjects take epitinib either once a day or twice a day. For twice a day epitinib uptake, on day 1/14/28, PK samples are collected predose, 1, 4, 8, 12 hours post-dose in the morning and 4 hours post-dose in the evening. On day 2/3/7, PK samples are collected predose, 4, 12 hours post-dose in the morning and 4 hours post-dose in the evening. On day 15/29/56, PK samples are collected predose in the morning.
  For once a day epitinib uptake, on day 1/14/28 PK samples are collected predose, 0.5, 1, 2, 4, 6, 8, 12 hours post-dose. On day 7, PK samples are collected predose and 4 hours post-dose. On day 2/15/29/56, PK samples are collected predose in the morning.

CONTACTS AND LOCATIONS:
Overall Officials: Rongjun Liu, M.D., Study Chair — Hutchison Medipharm Limited
Locations (1):
- Guangdong General Hospital, Guangzhou, China

REFERENCES:
- [Derived] Zhou Q, Wang M, Zhang H, Hong Q, Liu X, Lu P, Su W, Wu YL. Safety and Efficacy of Epitinib for EGFR-Mutant Non-Small Cell Lung Cancer With Brain Metastases: Open-Label Multicentre Dose-Expansion Phase Ib Study. Clin Lung Cancer. 2022 Sep;23(6):e353-e361. doi: 10.1016/j.cllc.2022.03.014. Epub 2022 May 7. PMID 35654732